CLINICAL TRIAL: NCT03916172
Title: Randomised Evaluation of Brief Psychological Intervention for Parents of Adolescents: The Open Door Approach to Parenting Teenagers (APT), in London, England
Brief Title: Evaluation of Psychological Intervention for Parents of Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Open Door Young People's Service (Other)
Responsible Party: Principal Investigator, Alex Desiatnikov, Dr. Alex Desiatnikov, Open Door Young People's Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 254697
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Parent-Child Relations
Keywords: Adolescence; Stress; Parent-adolescent relationship

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APT Treatment (Experimental): Participants in this arm will receive the Open Door Approach to Parenting Teenagers (APT). It offers 6 weekly 50-minute appointments with an optional 7th review session.
  Interventions: Behavioral: The Open Door Approach to Parenting Teenagers (APT)
- Waiting List (No Intervention): Participants in this group will be placed on a waiting list and will receive APT treatment after no longer than 25 weeks.

INTERVENTIONS:
Behavioral: The Open Door Approach to Parenting Teenagers (APT) — APT works on a one-to-one or couple basis. It offers 6 weekly 50-minute appointments with an optional 7th review session. The practitioners delivering the intervention have qualifications in psychology, or significant experience of working with adolescent populations, and have undertaken training and supervision in the model. Its aim is to help the parent manage the parenting of their teenager more effectively and establish a more balanced relationship by eliciting their views, feelings, and understanding of their teenager and their relationship, discussing their parental identity and role, carefully examining communication, responses, and information giving, and supporting appropriate boundary making. This is achieved through a collaborative development of strategies, psychoeducation and behavioural experiments.
  Arms: APT Treatment

SUMMARY:
Adolescence is a challenging period for young people and their parents. Changes during adolescence bring increases in social, psychological and behavioural problems (such as gang membership and drug abuse), and most long-lasting mental health problems start during this period. One of the strongest predictors of adolescent outcomes is the quality of parenting they receive at this stage. Parents often struggle with parenting adolescents, leading to feelings of stress and incompetence which, when reaching clinical levels, result in physical and mental health difficulties for parents and their children. This puts significant strain on community, social and mental health services. While the effectiveness of programmes to support parents of adolescents is certain, most are group-based and struggle to retain participants, especially amongst those who need help most: clinically stressed, and single parents. There are no standard care pathways for these parents, which leads to chronic problems and high long-term cost. The present study aims to measure the effectiveness of the Open Door's Approach to Parenting Teenagers (APT) - a manualised, six-session individual parenting intervention focusing on the relationship between parent and adolescent. This brief intervention, developed with awareness of the organisational realities and overarching aims of the National Health Service (NHS), has shown good results amongst clinically stressed parents in a pilot trial. The next phase in evaluating this approach is ruling out spontaneous recovery, by randomly assigning participants to APT or a waiting list control and comparing their results after the intervention, and again after 3 months. If successful, this study will have a major impact on communities around the United Kingdom (UK) - offering an evidence-based, non-proprietary intervention that can be easily disseminated.

DETAILED DESCRIPTION:
This study is the next step in the evaluation trajectory of the Open Door Approach to Parenting Teenagers (APT), and is a randomised controlled trial investigating whether receiving APT is more effective than being on a Waiting List (WL) in a sample of 60 parents of adolescents. We hypothesise that in comparison to those on the WL, those receiving APT will show significant improvements in:

* parental stress;
* parent-adolescent relationship;
* adolescent and parent wellbeing and mental health outcomes;

Secondary aims of the study will include:

* Ascertaining treatment fidelity
* Disseminating outcomes to inform policymakers, commissioners and providers, to facilitate evidence-based decisions about community services.

Procedure This trial will be carried out at two clinical sites in North London over 12months.

Method:

Parents and adolescents in the APT condition will be measured 3 times: at baseline, end-of-treatment, and follow-ups at three after the end-of-treatment. Those in WL will be measured three times from pre-treatment to three months follow-up. Then they will be offered APT. Measures are grouped into four batteries: for the parent, the adolescent, the therapist and an observer, and they will measure changes in parental stress, perceptions of the parent about their adolescent's psychopathology and relational problems, aspects of parenting relevant to aetiology and treatment of adolescent issues. The batteries also include variables mediating recovery, therapeutic alliance, health services utilisation and therapists' adherence to the ATP model.

Analysis plan:

The primary outcome will be analysed using within- and between-groups mean differences to estimate treatment effects. Results will be disseminated through scientific papers, academic conferences, the Open Door (OD) website, and reports will be distributed among educational and health institutions in our local network. If results have merit, the intervention manual will be published, and training will be offered to professionals outside OD. If successful, we anticipate this study to have a major impact on communities around the UK. It is a non-proprietary intervention that can be easily disseminated.

ELIGIBILITY:
Inclusion Criteria:

* Being a parent of an adolescent aged 11-18 years
* Adolescent currently lives with parent for a minimum of 2 days/week
* Parent demonstrates clinically significant levels of concern on primary measure (Stress Index for Parents of Adolescents)
* Parent must be proficient in English so they may fully understand the material presented to them during the research study

Exclusion Criteria:

* Parent currently receiving treatment for psychotic illness
* Parent previously received APT intervention
* Adolescent has severe developmental disorder (e.g. Autism Spectrum Disorder) or serious life threatening health impairment
* Adolescent currently receiving individual psychotherapeutic treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Stress Index for Parents of Adolescents (SIPA) | 5 months
  This is a 112-item, self report that is structured into three main domain scores: Adolescent Domain (AD), Parent Domain (PD), and Adolescent-Parent Relationship Domain (APRD). The AD has 4 subscale scores: Moodiness/Emotional Lability (MEL), Social Isolation/Withdrawal (ISO), Delinquency/Antisocial (DEL), and Failure to Achieve or Persevere (ACH). The PD also has 4 subscale: Life Restrictions (LFR), Relationship with Spouse/Partner (REL), Social Alienation (SOC) and Incompetence/Guilt (INC). The APRD has no subscales. The Index of Total Parenting Stress (TPS) is a composite score computed from all items. Scores are then classified into broad ranges: normal, borderline, clinically significant and clinically severe.

SECONDARY OUTCOMES:
Strengths And Difficulties Questionnaire Parent Version (SDQ-P) | 5 months
  Strengths and Difficulties Questionnaires (SDQ): a brief, parent-report, behavioural questionnaire. It comprises 25 items measuring emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behaviour. The measure has excellent psychometric properties, and national norms have been extracted from a large national survey of child and adolescent mental health carried out by the Office for National Statistics. For all time-points except baseline, a follow-up version of the measure will be used, which adds questions regarding the intervention's impact.
Strengths and Difficulties Questionnaire Young Person Version (SDQ-YP) | 5 Months
  Strengths and Difficulties Questionnaires (SDQ): a brief, self-report, behavioural questionnaire. It comprises 25 items measuring emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behaviour. The measure has excellent psychometric properties, and national norms have been extracted from a large national survey of child and adolescent mental health carried out by the Office for National Statistics. For all time-points except baseline, a follow-up version of the measure will be used, which adds questions regarding the intervention's impact.
Alabama Parenting Questionnaire - Short Form (APQ-SF) | 5 months
  A 12-item, self- report measure that focuses on parenting behaviours. The parent APQ measures five dimensions of parenting that are relevant to the aetiology and treatment of child and adolescent problems: positive involvement with children, supervision and monitoring, use of positive discipline techniques, consistency in the use of such discipline and use of corporal punishment. The APQ has good psychometric properties and has shown good discrimination between clinical and non-clinical groups.
Patient Health Questionnaire Module 9 (PHQ-9) | 5 months
  A screen for depression, extensively used in the literature and clinical practice, with excellent psychometric properties.
Generalised Anxiety Disorder Screener (GAD-7) | 5 months
  A 7-item screen with good sensitivity and specificity to capture and distinguish anxiety symptoms and disorders. Extensively used in clinical and research contexts.
Alabama Parenting Questionnaire Young Person version (APQ-YP) | 5 months
  This measure is complementary to the parent version described above. It measures adolescents' perceptions about the parenting they receive.
EQ-5D-5L | 5 months
  This is a standardised instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. It consists of a descriptive system and the EQ Visual Analogue Scale (VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
Reflective Function Questionnaire (RFQ) | 5 months
  A brief, easy-to-administer screening measure of reflective functioning. It comprises 8 items yielding two sub-scales assessing certainty and uncertainty of mental states.
Conflict Behaviour Questionnaire (CBQ) | 5 months
  A 20-item questionnaire that assesses perceived communication and conflict in the parent-adolescent relationship. The CBQ has good psychometric properties and has been found to successfully discriminate between distressed and non-distressed families. Both parent-report and self-report for adolescent versions will be used.
Parenting Scale (PS) | 5 months
  This is a 30-item questionnaires that measures two dysfunctional discipline styles in parents: Laxness and Over-reactivity, and also measures verbosity. This scale has good psychometric properties and has been found to discriminate between parents of clinic and non-clinic children.
Goal Based Measure | 5 months
  Developed by the Child Outcomes Research Consortium. Part of Open Door's regular practice. It is a simple form that lists the patient's goals for the treatment, and every session the patient rates their accomplishment from zero to ten.
Working Alliance Inventory-Short Form-Client (WAI-SF-C) | 5 months
  This measure will only be included in the end- of-treatment battery. This is a 12 item questionnaire , which assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. This brief measure has excellent psychometric properties.
Working Alliance Inventory-Short Form-Therapist (WAI-SF-T) | 5 months
  The therapist counterpart for the measure listed above. It will be completed by therapists at the end of treatment and is a 12-item scale that measures the alliance elements described above.
Working Alliance Inventory-Observer (WAI-O) | 5 months
  The observer counterpart of the measure described above. It is a 32-item scale that measures the alliance elements described above.
Experience of Services Questionnaire | 5 months
  This measure will only be included in the end-of-treatment battery. This is part of Open Door's regular practice. The questionnaire addresses the quality of service provided: how well the intervention met the participants' needs, increased their skills, decreased the adolescent's problem behaviours, and whether the participants would recommend the program to others.
Adherence to the APT Model | 5 months
  The APT manualised model includes checklists to be filled out by observers for each of the six sessions. Only 1 session per participant will be scored and scoring will be performed by supervisors on a randomly selected intervention session's video. These checklists contain both concrete actions the therapist must carry out during the selected session and elements regarding both the therapeutic stance, such as level of activity/passivity of the therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Desiatnikov, Principal Investigator — Open Door Young People's Consultation Service
Locations (1):
- Open Door Young People's Consultation Service, London, United Kingdom